CLINICAL TRIAL: NCT01244568
Title: Acceleration Adoption of Comparative Effectiveness Research Results With Patient Decision Support Intervention and Treatment- Study 2
Brief Title: Decision Support Interventions (DESI) for Prostate Cancer Screening and Treatment - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Palo Alto Medical Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Carmen Lewis, MD, MPH, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-1318; 1R18AE000023-01 (NIH)
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Decision support interventions (DESI); Comparative Effectiveness Research (CER)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- Prostate cancer treatment DESI (Experimental)
  Interventions: Behavioral: Prostate cancer treatment DESI

INTERVENTIONS:
Behavioral: Prostate cancer treatment DESI — DESI is a 50 minute program on treatment choices for prostate cancer that will be given out to the experimental group. The program explains several treatment options including surgery (radical prostatectomy), radiation therapy (external beam and/or brachytherapy), hormone therapy, and active surveillance and watchful waiting. The program's intended audience is men with early state prostate cancer who are trying to make a treatment decision.
  Other Names: Decision Support Intervention
  Arms: Prostate cancer treatment DESI

SUMMARY:
Researchers in this study will determine whether providing decision support interventions (DESIs) to men with low risk prostate cancer improves their decision-specific knowledge and alters their treatment decisions.

DETAILED DESCRIPTION:
Potentially eligible men (age 45 and older who have localized prostate cancer with a Gleason score of 6 or less) will be identified and recruited to participate in the study before their next office visit. Patients who are interested and provide informed consent will be asked to complete a brief survey about background, medical history, knowledge of prostate cancer and health-related quality of life. Once the survey is completed the patient will be randomly assigned to one of 2 groups. Those assigned to the "Usual Care" group will not receive any additional information materials as part of their participation in the study. Those assigned to the "Patient Decision Support" group will receive a DVD program that contains information about treatment choices for prostate cancer.

Participants will be asked to answer a brief telephone survey at 3 and 6 months from the day of their last office visit. Survey questions will ask about knowledge about prostate cancer, health-related quality of life, whether or not the DVD was viewed and what treatment decision was made.

Research staff will also review medical records 6 months after enrollment to determine which treatment was received for prostate cancer, how many visits with health care providers were completed since enrollment and which medical services and procedures were received.

ELIGIBILITY:
Inclusion Criteria:

Age 45 or older Localized prostate cancer with a Gleason score of 6 or less

Exclusion Criteria:

Women

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Active treatment vs. Watchful waiting/active surveillance at 3 and 6 months | 3 and 6 month follow-up
  Men who review a DESI before making a treatment decision will be more likely to choose active surveillance/watchful waiting and will have better decision-specific knowledge.

SECONDARY OUTCOMES:
DESI viewing | 3 month follow-up (phone survey)
  Decision aid viewing is a self-reported measures. Patients will be asked if they viewed the DVD that was given to them (intervention group)prior to them making a treatment choice decision.
Healthcare utilization | 6 month follow-up
  Research staff will review EMR data to access decision-making outcomes and resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen L Lewis, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Ming Tai-Seale, Ph.D, MPH, Principal Investigator — Palo Alto Medical Foundation
Locations (2):
- United States (2):
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina